CLINICAL TRIAL: NCT02196870
Title: Physiological Effects of Chest Wall Elastance on Pulmonary Mechanics of Acute Respiratory Failure Patientstranspulmonary Pressure
Brief Title: Effects of Chest Wall Elastance on Pulmonary Mechanics of Acute Respiratory Failure (ARF)
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Department of Critical Care Medicine, Zhong-Da Hospital, Southeast University, China
Other Study IDs: Chest wall Elastance in ARF
Record Dates: First submitted 2014-07-12; First posted 2014-07-22 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Airway Pressure Stress Index; Transpulmonary Pressure Stress Index; Acute Respiratory Failure; Chest Wall Elastance
Keywords: Airway pressure stress index; Transpulmonary pressure stress index; Acute Respiratory Failure; Chest wall elastance; Lung stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with chest wall elastance increasing could worsen lung function. Increasing of chest wall elastance plays a great role in lung mechanics, and could influence mechanical ventilation settings. Therefore, It could help the physicians to find appropriate indicators and optimize the treatments of ARF patients to explore the mechanisms of lung mechanics changse in the patients with high chest wall elastance.

DETAILED DESCRIPTION:
Mechanical ventilation(MV) is an important treatment for acute respiratory failure(ARF) patients, could improve hypoxemia, maintain lung volume and promote alveolar opening. However, because of barotrauma, volutrauma and biotrauma, MV could cause or aggravate acute lung injury not only in acute respiratory distress syndrome(ARDS) patients, but in patients with normal lung function1,2.

Patients with chest wall elastance increasing could worsen lung function. Increasing of chest wall elastance plays a great role in lung mechanics, and could influence mechanical ventilation settings. Therefore, It could help the physicians to find appropriate indicators and optimize the treatments of ARF patients to explore the mechanisms of lung mechanics changse in the patients with high chest wall elastance.

The present study is set out to examine the effects of high chest wall elastance on changes of lung mechanics and the correlation of airway pressure(Paw) stress index and transpulmonary pressure(PL) stress index.

ELIGIBILITY:
Inclusion Criteria:

* ARF
* mechanical ventilation
* cardiovascular stable

Exclusion Criteria:

* age < 18y or > 85y
* pregnancy
* COPD or chronic pulmonary disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute respiratory failure patients
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes of oxygenation and lung mechanics | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Xie, Dr., Principal Investigator — Zhongda hospital, Southeast University, Jiangsu, China
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Pan C, Chen L, Zhang YH, Liu W, Urbino R, Ranieri VM, Qiu HB, Yang Y. Physiological Correlation of Airway Pressure and Transpulmonary Pressure Stress Index on Respiratory Mechanics in Acute Respiratory Failure. Chin Med J (Engl). 2016 Jul 20;129(14):1652-7. doi: 10.4103/0366-6999.185855. PMID 27411451